CLINICAL TRIAL: NCT07006064
Title: Comparison of SuperNO₂VA™ Nasal Mask and Conventional Nasal Oxygen Therapy in Preventing Hypoxia During Sedation for TAVI Procedures in Geriatric Patients
Brief Title: Preventing Hypoxia in Sedated TAVI: SuperNO₂VA vs. Conventional Oxygen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Bilkent Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Muhammed Talha Daşgın, Anesthesiology and Reanimation Doctor, Principal Investigator, Ankara Bilkent Sehir Hastanesi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ankara Bilkent City Hospital; Muhammed Talha (Other: Ankara Bilkent City Hospital)
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; Transcatheter Aortic Valve Implantation (TAVI); hypoxia; SuperNO 2 VA™ mask; end-tidal CO2
MeSH Terms: conditions — Aortic Valve Stenosis; Hypoxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SUPERNOVA MASK (Active Comparator)
  Interventions: Device: SUPERNOVA
- NASAL MASK (Active Comparator)
  Interventions: Device: NASAL MASK

INTERVENTIONS:
Device: SUPERNOVA — In the intervention group, oxygen is delivered using the SuperNO2VA™ nasal positive airway pressure mask (Vyaire Medical, USA), which differs from conventional nasal oxygen delivery systems by providing continuous positive airway pressure (CPAP) through a sealed nasal interface. This mask also includes an integrated sampling port for accurate end tidal carbon dioxide (EtCO2) monitoring. The aim is to reduce the incidence of hypoxia and allow for better detection and prevention of hypo/hypercapnia during sedation in elderly patients undergoing TAVI without intubation. The use of positive pressure is intended to prevent upper airway collapse, maintain functional residual capacity, and improve gas exchange during sedation.
  Arms: SUPERNOVA MASK
Device: NASAL MASK — Traditional nasal cannulas only provide passive oxygen flow. End-tidal CO2 measurement is being conducted with Capnostream™ 35 Portable Respiratory Monitor.
  Arms: NASAL MASK

SUMMARY:
With increasing life expectancy, the geriatric population continues to grow. According to the Turkish Statistical Institute (TÜİK), the average life expectancy in Turkey between 2021 and 2023 is 77.3 years. As the number of elderly surgical patients rises, optimizing anesthesia care is critical to reducing complications and improving clinical outcomes. In elderly patients with severe aortic stenosis, traditional surgical aortic valve replacement poses a high risk of complications. Consequently, Transcatheter Aortic Valve Implantation (TAVI) has emerged as a preferred, less invasive alternative. Due to technological advancements and shorter procedure durations, TAVI is increasingly performed under sedation rather than general anesthesia. However, sedation carries risks, including hypoxemia and hypoventilation, primarily due to sedative-induced respiratory depression.

Pulse oximetry, the traditional monitoring method, measures only peripheral oxygen saturation and does not provide early detection of apnea or hypoventilation. Therefore, monitoring end-tidal carbon dioxide (EtCO₂) during sedation has gained importance. The American Society of Anesthesiologists (ASA) recommends EtCO₂ monitoring during sedation. However, obtaining accurate EtCO₂ values via nasal cannulas is technically challenging. Open sampling ports and high oxygen flow rates can cause dilution or loss of exhaled CO₂, resulting in inaccurate readings.

The SuperNO₂VA™ nasal mask (Vyaire Medical, USA) addresses these limitations with an integrated CO₂ sampling port and the ability to provide positive airway pressure. This facilitates more accurate EtCO₂ monitoring and better ventilatory support compared to standard nasal cannulas. Prior studies have demonstrated that the SuperNO₂VA mask significantly reduces the risk and severity of hypoxia in high-risk patients during sedated endoscopic procedures. It prevents upper airway collapse and increases ventilated lung surface area, without causing clinically significant hypercapnia or CO₂ retention.

This study aims to compare the incidence of hypoxia in patients aged 65 years and older undergoing TAVI under sedation using either the SuperNO₂VA nasal mask or a conventional nasal oxygen mask. Secondary outcomes include the evaluation of intraoperative hypercapnia or hypocapnia and the assessment of postoperative respiratory complications.

DETAILED DESCRIPTION:
The continuous increase in life expectancy has led to steady growth in the geriatric population. According to the Turkish Statistical Institute (TÜİK), the average life expectancy in Turkey from 2021 to 2023 is 77.3 years. In surgical geriatric patients, optimizing anesthesia care strategies is essential to reduce complications and enhance clinical outcomes. In patients with severe aortic stenosis, traditional surgical aortic valve replacement is associated with a high risk of complications. As a result, Transcatheter Aortic Valve Implantation (TAVI) has gained popularity. The anesthetic approach to TAVI varies based on surgical preference, procedural volume, echocardiography type, and team experience. Recent technological advancements and shorter procedural durations have made sedation-based anesthesia a preferred option. However, sedation may result in complications such as hypoxemia and hypoventilation due to central respiratory depression from sedative agents. Pulse oximetry, a conventional respiratory monitoring method, measures only peripheral oxygen saturation and may delay the detection of hypoventilation or apnea. In sedated patients receiving supplemental oxygen, measuring exhaled carbon dioxide (CO2) becomes essential. The American Society of Anesthesiologists (ASA) has endorsed the use of end-tidal capnography (EtCO2) as a standard for monitoring sedation. While capnography surpasses pulse oximetry in detecting hypoventilation and apnea, accurate EtCO2 measurement during deep sedation remains technically challenging due to dilution of exhaled gases from open nasal cannula sampling ports and high oxygen flow rates. The SuperNO2VA™ nasal mask (Vyaire Medical, USA) is an innovative device designed to overcome these challenges. It features an integrated CO2 sampling port and provides positive airway pressure, thereby allowing for accurate EtCO2 measurement and improved respiratory support compared to standard nasal oxygen masks. Prior research has shown that the SuperNO2VA mask significantly reduces both the frequency and severity of hypoxia in high-risk patients undergoing sedated endoscopic procedures. This device also helps prevent upper airway collapse and enhances lung ventilation. Importantly, its use has not been associated with clinically significant hypercapnia or CO2 retention. The objective of this study is to compare the incidence of hypoxia in patients over 65 years of age undergoing TAVI under sedation, using either the SuperNO2VA nasal mask or a standard nasal oxygen mask. In minimally invasive procedures such as TAVI in the geriatric population, accurate evaluation of hypoxia and hypercapnia is critical. Traditional oxygen delivery methods may be insufficient in preventing hypoxia and predicting CO2 disturbances. Based on previous studies, it is hypothesized that the SuperNO2VA mask will reduce hypoxia and improve detection of hypo/ hypercapnia via continuous EtCO2 monitoring. No specific risk is anticipated for participants in this study. A prospective, randomized controlled trial is planned, enrolling 100 patients via computer generated randomization in a 1:1 ratio (SuperNO2VA group: 50; control group: 50). In patients undergoing TAVI under sedation without endotracheal intubation, the SuperNO2VA group will receive oxygen via the nasal mask delivering positive airway pressure, while the control group will receive oxygen through a standard nasal mask. Oxygen flow will be adjusted to maintain SpO2

* 92%. All parameters will be prospectively recorded by the clinical staff and investigators from the Department of Anesthesiology and Reanimation at Ankara Bilkent City Hospital. Study participation will be terminated for any patient in the event of withdrawal, intraoperative intubation, or serious adverse events such as laryngospasm. This study will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines. Written informed consent will be obtained from all participants, who will retain the right to withdraw from the study at any time without providing a reason.

Preoperative parameters to be assessed:

Age and sex Height, weight, Body Mass Index (BMI) ASA Physical Status Classification Comorbidity evaluation Smoking history ARISCAT score parameters

Intraoperative parameters to be assessed:

Duration of anesthesia Occurrence of complications (e.g., need for intubation, resuscitation, bronchospasm) Incidence of hypoxia (SpO2 < 90% for >10 seconds) Continuous EtCO2 monitoring Arterial blood gas measurements (PaO2, PaCO2) Peripheral oxygen saturation (SpO2) will be monitored continuously and recorded throughout the preoperative, intraoperative, and postoperative periods, totaling 12 hours. Data will be analyzed using SPSS version 27 (IBM Corporation, Armonk, NY, USA). Descriptive statistics will summarize baseline characteristics. The incidence of hypoxia between groups will be compared using Fisher's Exact Test. Multivariate logistic regression will be used to identify factors associated with hypoxia or hypercapnia. Statistical significance will be defined as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older who are scheduled for TAVI under sedation will be included in the study.

Exclusion Criteria:

* History of prolonged intubation
* History of tracheostomy
* Patients who are planned to undergo endotracheal intubation during the procedure
* Patients undergoing TAVI under local anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Hypoxia (SpO₂ < 90% for >10 Seconds) | 12 hours
  Each patient included in the study will be monitored noninvasively with a pulse oximeter for oxygen saturation when taken to the operating room. The pulse oximeter will be placed on the index finger of the right hand. Oxygen saturation will be recorded as a numerical value between 0-100. Values below 90 will be evaluated as hypoxia and intervention will be made. Values below 90 will be evaluated as hypoxia and appropriate intervention will be made. A drop in SpO₂ below 90% lasting longer than 10 seconds will be recorded as hypoxia.

SECONDARY OUTCOMES:
Number of Participants with Hypotension (MAP < 65 mmHg | 12 hours
  Each patient included in the study will be noninvasively monitored for arterial blood pressure upon arrival in the operating room. A standard noninvasive blood pressure cuff will be placed on the left upper arm. Arterial blood pressure values will be recorded in mmHg as systolic, diastolic, and mean arterial pressure (MAP). A MAP value below 65 mmHg will be considered hypotension, and appropriate intervention will be performed.
Number of Participants with Hypoxemia (PaO2 < 60 mmHg) | 12 hours
  Following the modified Allen test, arterial cannulation will be performed primarily from the radial artery under ultrasound guidance. Arterial blood gas analysis will be performed intraoperatively. The arterial partial pressure of oxygen (PaO2) will be measured and recorded in mmHg. A PaO2 value below 60 mmHg will be considered significant hypoxemia, and appropriate interventions will be undertaken.
Number of Participants with Hypercapnia or Hypocapnia (PaCO2 > 45 or < 35 mmHg) | 12 hours
  Following the modified Allen test, arterial cannulation will be performed primarily from the radial artery under ultrasound guidance.Arterial blood gas analysis will also include the measurement of arterial partial pressure of carbon dioxide (PaCO2). Values will be recorded in mmHg. A PaCO2 level above 45 mmHg will be interpreted as hypercapnia, while values below 35 mmHg will indicate hypocapnia. Clinical interventions will be made accordingly.
Mean and Abnormal EtCO2 Levels During Sedation (EtCO2 < 30 or > 50 mmHg) | 12 hours
  End-tidal carbon dioxide (EtCO2) monitoring will be performed continuously throughout the intraoperative period using a capnograph connected to the anesthesia circuit. EtCO2 values will be recorded in mmHg. Values outside the normal physiological range (35-45 mmHg) will be evaluated in the context of ventilation status. EtCO2 < 30 mmHg will be considered as hypocapnia, while EtCO2 > 50 mmHg will be interpreted as hypercapnia, and necessary interventions will be carried out.
Number of Participants Experiencing Intraoperative Complications (Intubation, Resuscitation, or Bronchospasm) | 12 hours
  Intraoperative complications will be evaluated and recorded. These include the need for endotracheal intubation, the need for resuscitation, and the occurrence of bronchospasm. Each event will be documented with its timing and clinical context. All interventions performed in response to these complications will also be recorded in detail. Patients who develop any of these complications intraoperatively will be excluded from the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedro, M. and Cataldo, S. (2020) Validation of Novel Completely Sealed Nasal Positive Airway Pressure Device: SuperNO 2 VA™ EtCO 2 Measurement and Pressure Test Performance. Open Journal of Anesthesiology, 10, 337-348. doi: 10.4236/ojanes.2020.1010030 .
- [Background] Kalner A, Kuchler F, Kavallari E, Muller M, Seufferlein T, Walter BM. Efficiency and safety of nasal positive airway pressure systems during endoscopic procedures in high-risk patients: Endo-Breath study. Endosc Int Open. 2024 May 29;12(5):E704-E714. doi: 10.1055/a-2306-9144. eCollection 2024 May. PMID 38812697
- [Background] Luzzi C, Orlov D, Foley K, Horlick E, Osten M, Cusimano RJ, Djaiani G. Choice of anesthesia technique is associated with earlier hospital discharge and reduced costs after transcatheter transfemoral aortic valve implantation. J Thorac Dis. 2024 Mar 29;16(3):1836-1842. doi: 10.21037/jtd-23-1739. Epub 2024 Mar 27. PMID 38617787
- See also: Related Info — https://data.tuik.gov.tr/Bulten/Index?p=Hayat-Tablolari-2021-2023-53678